CLINICAL TRIAL: NCT06049225
Title: Medical Nutrition Therapy and Diabetes Self-Management Education for People With Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-300010728; SBIR-PHASE2 (Other: Kamin Consulting Inc)
Record Dates: First submitted 2023-08-24; First posted 2023-09-22 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Physical Disability
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: High-Tech Intervention Group (Experimental): Those in the high-tech intervention group will receive 6 months of active intervention (up to 60 minutes weekly health coaching calls and content delivery) and technology access.
  Interventions: Behavioral: High-Tech
- Experimental: Low-Tech Intervention Group (Experimental): Those in low-tech group will receive 6 months of one weekly coaching calls (last up to 60 minutes) and one weekly email
  Interventions: Behavioral: Low-Tech
- Active Comparator: Attention Control Group (Active Comparator): The control group will be used to provide an untreated comparison for the intervention groups and will not receive MNT or technology support. Participants in the control arm will only get a baseline and post-intervention testing.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: High-Tech — Access to technological platform and weekly health coaching
  Arms: Experimental: High-Tech Intervention Group
Behavioral: Low-Tech — Weekly email with educational content and weekly health coaching
  Arms: Experimental: Low-Tech Intervention Group
Behavioral: Attention Control — No technology access or health coaching
  Arms: Active Comparator: Attention Control Group

SUMMARY:
The purpose of this project is to develop, and pilot test an accessible and inclusive medical nutrition therapy and diabetes self-management education program for people with Type 2 Diabetes and physical disabilities.

DETAILED DESCRIPTION:
This study will use a three-arm randomized control trial design. Eligible and consented participants will be assigned to one of three groups: (1) intervention with high-tech support, (2) intervention with low-tech support, and (3) attention-control group. The active intervention period will include six months of weekly health coaching calls and technology access. The low-tech support group will receive six months of weekly coaching calls and weekly email containing related materials in PDF format but no video and technology content.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of T2DM
2. 18 to 65 years of age
3. Living with a permanent physical disability such as SCI, spina bifida, multiple sclerosis, stroke
4. Ability to converse in and read English
5. Availability of a smartphone or computer that can run apps
6. Have internet connection capabilities

Exclusion Criteria:

1. Current enrollment in any diabetes related intervention
2. Present or soon-planned pregnancy
3. Major heart attack or heart surgery in the past 12 months
4. Have undergone a dialysis, kidney transplant or a kidney surgery in the past 12 months
5. Severe cognitive impairment
6. Severe untreated depression in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Diabetes Quality of Life | 24 weeks
  Measured using the DQoL (Diabetes Quality of Life Measure) Questionnaire; Minimum score =1; maximum score = 5; Higher score represents worse outcome
Psychological Distress | 234 weeks
  Measured using Diabetes Distress Scale (DDS); Minimum score = 1, maximum score = 6; Higher score represents worse outcome
Self-efficacy | 24 weeks
  Measured using Diabetes Empowerment Scale; Minimum score = 1; maximum score = 5; Higher score represents better outcome

SECONDARY OUTCOMES:
Glycemic Management | 24 weeks
  Measured using HbA1c

OTHER OUTCOMES:
Physical Activity | 24 weeks
  Measured using Godin leisure-time exercise questionnaire; Minimum score = 0; Maximum score = unknown; Higher score represents better outcome
Dietary intake | 24 weeks
  Measured using The US version of the Diabetes and Diet Questionnaire
Medication Adherence | 24 weeks
  Measured using the Medication Adherence Rating Scale
Health Dashboard Usability | 24 weeks
  Measured using the System Usability Scale; Maximum item score (Strongly agree) = 5, minimum item score (Strongly disagree) = 1; Higher scores represent better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. Economic Costs of Diabetes in the U.S. in 2017. Diabetes Care. 2018 May;41(5):917-928. doi: 10.2337/dci18-0007. Epub 2018 Mar 22. PMID 29567642
- [Background] Hall L, Colantonio A, Yoshida K. Barriers to nutrition as a health promotion practice for women with disabilities. Int J Rehabil Res. 2003 Sep;26(3):245-7. doi: 10.1097/00004356-200309000-00013. PMID 14501578
- [Background] Kayes NM, Schluter PJ, McPherson KM, Taylor D, Kolt GS. The Physical Activity and Disability Survey -- Revised (PADS-R): an evaluation of a measure of physical activity in people with chronic neurological conditions. Clin Rehabil. 2009 Jun;23(6):534-43. doi: 10.1177/0269215508101750. Epub 2009 May 15. PMID 19447843
- [Derived] Aboagye A, Peckham J, Hearld KR, Abdullah S, Thirumalai M. A Technology-Enhanced Medical Nutrition Therapy and Diabetes Self-Management Education for Adults With Disability and Type 2 Diabetes: Protocol for a Pilot and Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 26;14:e71495. doi: 10.2196/71495. PMID 41002071